CLINICAL TRIAL: NCT02124785
Title: Long-term Persistence of Hepatitis A Antibodies in Healthy Adults, Primed 21 to 25 Years Earlier With GSK Biologicals' Hepatitis A Vaccine Havrix® (SB208109) in Studies HAV-112 (208109/108) or HAV-123 (208109/114)
Brief Title: Evaluation of the Long-term Persistence of Hepatitis A Antibodies in Healthy Adults Who Were Vaccinated 21-25 Years Earlier With GlaxoSmithKline (GSK) Biologicals' Hepatitis A Vaccine, Havrix®
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: This study has been cancelled before initiation due to company's prioritisation decisions linked to resources restrictions.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 116763; 2013-001918-15 (EudraCT Number)
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Hepatitis A
Keywords: Long-term persistence; Havrix; Hepatitis A
MeSH Terms: conditions — Hepatitis A | interventions — Blood Specimen Collection

ARMS (1):
- HAV Group (Experimental): Subjects who were previously vaccinated with Havrix in primary studies.
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — At Years 21 to 25 after their second vaccine dose.

SUMMARY:
The purpose of this study is to assess the long-term persistence of immunity to hepatitis A in adults who were vaccinated 21-25 years earlier with hepatitis A vaccine, Havrix®.

DETAILED DESCRIPTION:
This is a long-term persistence study in which subjects who participated in the primary studies HAV-112 (208109/108) or HAV-123 (208109/114) and did not receive an additional dose of hepatitis A vaccine since then, will be invited to provide a blood sample at Years 21 to 25 after their second vaccine dose. No vaccine will be administered during the study period.

ELIGIBILITY:
Inclusion Criteria:

* A male or female who received two doses of Havrix in study HAV-112 (208109/108) or HAV-123 (208109/114), and received no further booster dose since then.
* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g. return for follow-up visits).
* Written informed consent obtained from the subject.

Exclusion Criteria:

* History of hepatitis A disease since completion of the primary vaccination series in studies HAV-112 (208109/108) or HAV-123 (208109/114).
* Administration of a hepatitis A vaccine at any time since completion of the primary vaccination series in studies HAV-112 (208109/108) or HAV-123 (208109/114) including a challenge dose of the study vaccine, as a part of the study procedures, during the long-term persistence phase.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history.
* Administration of hepatitis A immunoglobulins and/or any blood products and/or long-acting immune-modifying drugs within six months prior to study entry.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to study entry. For corticosteroids, this will mean prednisone ≥ 20 mg/day, or equivalent. Inhaled and topical steroids are allowed.
* Administration of long-acting immune-modifying drugs within six months prior to study entry (e.g. infliximab).
* Concurrently participating in another clinical study during the period starting 30 days before and ending 30 days after each study visit, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity with respect to components of the study vaccine in terms of anti-HAV seropositivity status and GMCs. | 21 to 25 years after the second vaccine dose.

SECONDARY OUTCOMES:
Occurrence of serious adverse events (SAEs). | During the entire study period (Year 21 to Year 25).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wilrijk, Belgium